CLINICAL TRIAL: NCT04773522
Title: A Phase 1 Study of JNJ-64407564, a Humanized GPRC5D * CD3 Bispecific Antibody in Japanese Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of JNJ-64407564 in Japanese Participants With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108930; 64407564MMY1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-02-25; First posted 2021-02-26 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — talquetamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Talquetamab (Experimental): Participants will receive talquetamab injection subcutaneously (SC) in 3 cohorts: Cohort 1 and Cohort 2 as 2 step-up doses and Cohort 3 as 3 step-up doses followed by a treatment dose.
  Interventions: Drug: Talquetamab

INTERVENTIONS:
Drug: Talquetamab — Talquetamab will be administered subcutaneously.
  Other Names: JNJ-64407564

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability in Japanese participants with relapsed or refractory multiple myeloma (MM) at the recommended Phase 2 dose (RP2D) identified in NCT03399799 study.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of multiple myeloma according to International Myeloma Working Group (IMWG) diagnostic criteria
* Participants must be relapsed or refractory to established therapies with known clinical benefit in relapsed/refractory multiple myeloma (MM) or be intolerant of those established MM therapies, and a candidate for talquetamab treatment in the opinion of the treating physician. Prior lines of therapy must include a proteasome inhibitor (PI), an immunomodulatory drug (IMiD) and an anti-CD38 antibody in any order during the course of treatment. Participants who could not tolerate a PI, immunomodulatory drugs or anti-CD38 antibody are allowed
* Eastern cooperative oncology group (ECOG) performance status grade of 0 or 1 at screening and immediately before the start of study treatment administration
* Women of childbearing potential must have a negative pregnancy test at screening and within 24 hours prior to the first dose of study treatment using highly sensitive pregnancy test either serum (Beta-human chorionic gonadotropin [Beta-hCG]) or urine
* Participants (or a legally acceptable representative) must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study. Consent is to be obtained prior to the initiation of any study-related tests or procedures that are not part of standard-of-care for the participant's disease

Exclusion Criteria:

* Toxicities from previous anticancer therapies that have not resolved to baseline levels or to Grade 1 or less except for alopecia or peripheral neuropathy
* Received a cumulative dose of corticosteroids equivalent to >=140 milligrams (mg) of prednisone within the 14-day period before the first step-up dose of study treatment (does not include pretreatment medication)
* Central nervous system involvement or clinical signs of meningeal involvement of multiple myeloma. If either is suspected, whole brain magnetic resonance imaging (MRI) and lumbar cytology are required during screening
* Pulmonary compromise requiring supplemental oxygen use to maintain adequate oxygenation
* Known allergies, hypersensitivity, or intolerance to the excipients of talquetamab

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to 1.5 years
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study.
Number of Participants With Serious Adverse Events (SAEs) | Up to 1.5 years
  A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Cohorts 1 and 2: Number of Participants With Dose-Limiting Toxicity (DLT) | Up to 28 days
  Number of participants with DLT will be reported. The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.
Cohort 3: Number of Participants With DLT | Up to 38 days
  Number of participants with DLT will be reported. The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.

SECONDARY OUTCOMES:
Serum Concentrations of JNJ-64407564 | Up to 1.5 years
  Serum concentrations of JNJ-64407564 will be assessed.
Systemic Cytokine Concentrations | Up to 1.5 years
  Cytokine concentrations such as concentration of interleukin (IL)-6, Interferon (IFN)-gamma, IL-10 and IL-2 receptors will be measured for biomarker assessment.
Number of Participants With Anti-Talquetamab Antibodies | Up to 1.5 years
  Number of participants with anti-talquetamab antibodies will be reported for immunogenicity assessment.
Number of Participants With Objective Response | Up to 1.5 years
  Objective response is defined as the participants with a partial response (PR) or better according to the International Myeloma Working Group (IMWG) criteria.
Duration of Response (DOR) | Up to 1.5 years
  DOR is defined as the duration from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the IMWG criteria, or death.
Time to Response (TTR) | Up to 1.5 years
  TTR is defined as the time between date of first dose of study treatment and the first efficacy evaluation that the participant has met all criteria for PR or better.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (6):
- Japan (6):
  - Shonan Kamakura General Hospital, Kamakura-shi
  - National Cancer Center Hospital East, Kashiwa
  - Nagoya City University Hospital, Nagoya
  - National Hospital Organization Okayama Medical Center, Okayama
  - Japanese Red Cross Medical Center, Shibuya City
  - Iwate Medical University Hospital, Shiwa-gun

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency